CLINICAL TRIAL: NCT00169442
Title: Immune Memory of GSK's DTPw-HBV/Hib Vaccine by Giving Plain PRP Polysaccharide at 10 Mths. Immuno & Reacto of a Booster Dose of DTPw-HBV/Hib or DTPw-HBV or DTPw-HBV+Hib at 15-18 Mths in Infants Previously Primed With DTPw-HBV/Hib
Brief Title: Immune Memory of DTPw-HBV/Hib Vaccine Following Primary Vaccination, Immuno & Reacto of a Booster Dose Given in Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 104065
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2017-02-28 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2017-05

CONDITIONS: Whole Cell Pertussis; Diphtheria; Hepatitis B; Tetanus; Haemophilus Influenzae Type b
MeSH Terms: conditions — Diphtheria; Hepatitis B; Tetanus; Haemophilus Infections | interventions — Hiberix; Vaccines

ARMS (6):
- Tritanrix-HepB/Hiberix Kft. Mix Group (Experimental): Healthy male and female infants who were primed with Tritanrix™-HepB/Hiberix™ Kft. vaccine, received a booster dose of Tritanrix™-HepB/Hiberix™ Kft. administered intramuscularly into the right upper thigh, at 15-18 months of age.
  Interventions: Biological: Tritanrix™-HepB/Hiberix™ Kft.
- Tritanrix-HepB/Hiberix Kft. Ref Group (Experimental): Healthy male and female infants who were primed with Tritanrix™-HepB/Hiberix™ vaccine, received a booster dose of Tritanrix™-HepB/Hiberix™ Kft. administered intramuscularly into the right upper thigh, at 15-18 months of age.
  Interventions: Biological: Tritanrix™-HepB/Hiberix™ Kft.; Biological: Tritanrix™-HepB/Hiberix™
- HB Tritanrix-HepB/Hiberix Kft. Mix Group (Experimental): Healthy male and female infants who were primed with Tritanrix™-HepB/Hiberix™ Kft. vaccine (with HepB at birth), received a booster dose of Tritanrix™-HepB/Hiberix™ Kft. administered intramuscularly into the right upper thigh, at 15-18 months of age.
  Interventions: Biological: Tritanrix™-HepB/Hiberix™ Kft.
- Tritanrix-HepB Kft.+Hiberix Group (Experimental): Healthy male and female infants who were primed with Tritanrix™-HepB Kft. and Hiberix™ vaccines, were boosted with Tritanrix™-HepB Kft. vaccine administered intramuscularly into the right upper thigh and Hiberix™ vaccine, administered intramuscularly into the left upper thigh, at 15-18 months of age.
  Interventions: Biological: Hiberix™; Biological: Tritanrix™-HepB Kft
- PRP Tritanrix-HepB Kft. Mix Group (Experimental): Healthy male and female infants who were primed with Tritanrix™-HepB/Hiberix™ Kft. vaccine, received plain Polyribosil-Ribitol-Phosphate (PRP) polysaccharide vaccine administered intramuscularly into the right upper thigh, at 10 months of age, followed by a booster dose of Tritanrix™-HepB Kft. administered intramuscularly into the right upper thigh, at 15-18 months of age.
  Interventions: Biological: Tritanrix™-HepB/Hiberix™ Kft.; Biological: Polyribosil-Ribitol-Phosphate (PRP) vaccine; Biological: Tritanrix™-HepB Kft
- PRP Tritanrix-HepB Kft. Ref Group (Experimental): Healthy male and female infants who were primed with Tritanrix™-HepB/Hiberix™ vaccine, received plain Polyribosil-Ribitol-Phosphate (PRP) polysaccharide vaccine administered intramuscularly into the right upper thigh, at 10 months of age, followed by a booster dose of Tritanrix™-HepB Kft. administered intramuscularly into the right upper thigh, at 15-18 months of age.
  Interventions: Biological: Tritanrix™-HepB/Hiberix™; Biological: Polyribosil-Ribitol-Phosphate (PRP) vaccine; Biological: Tritanrix™-HepB Kft

INTERVENTIONS:
Biological: Tritanrix™-HepB/Hiberix™ Kft. — GlaxoSmithKline (GSK) Biologicals Korlatolt Felelossegu Tarsasag [Kft] (Limited Company) combined diphtheria (D), tetanus (T), whole cell Bordetella pertussis (Pw), hepatitis B vaccine with new sources of D, T and Pw antigens mixed with Haemophilus influenzae type b (Hib2.5) vaccine.
  Other Names: DTPw-HBV/Hib Kft
  Arms: HB Tritanrix-HepB/Hiberix Kft. Mix Group; PRP Tritanrix-HepB Kft. Mix Group; Tritanrix-HepB/Hiberix Kft. Mix Group; Tritanrix-HepB/Hiberix Kft. Ref Group
Biological: Tritanrix™-HepB/Hiberix™ — GSK Biologicals' combined diphtheria, tetanus, whole cell Bordetella pertussis, hepatitis B and Haemophilus Influenzae type b vaccine
  Other Names: DTPw-HBV/Hib
  Arms: PRP Tritanrix-HepB Kft. Ref Group; Tritanrix-HepB/Hiberix Kft. Ref Group
Biological: Hiberix™ — GSK Biologicals' Haemophilus influenzae type b vaccine
  Arms: Tritanrix-HepB Kft.+Hiberix Group
Biological: Polyribosil-Ribitol-Phosphate (PRP) vaccine — plain PRP polysaccharide vaccine
  Arms: PRP Tritanrix-HepB Kft. Mix Group; PRP Tritanrix-HepB Kft. Ref Group
Biological: Tritanrix™-HepB Kft — GSK Biologicals Korlatolt Felelossegu Tarsasag [Kft] (Limited Company) combined diphtheria, tetanus, whole cell Bordetella pertussis, hepatitis B vaccine with new sources of D, T and Pw antigens produced at GSK Biologicals Kft., Gödöllö, Hungary.
  Other Names: DTPw-HBV Kft
  Arms: PRP Tritanrix-HepB Kft. Mix Group; PRP Tritanrix-HepB Kft. Ref Group; Tritanrix-HepB Kft.+Hiberix Group

SUMMARY:
To assess the immune memory following primary vaccination of DTPw-HBV/Hib vaccine and to assess immunogenicity and reactogenicity of a booster dose given at 15 - 18 months of age.

DETAILED DESCRIPTION:
* Subjects who received DTPw-HBV/Hib in the primary vaccination without HBV at birth will be randomised (1:3 ratio) to receive either: Plain PRP at 10 months of age followed by DTPw-HBV at 15-18 months of age or DTPw-HBV/Hib at 15-18 months of age.
* Subjects who received DTPw-HBV + Hib in the primary vaccination without HBV at birth will receive DTPw-HBV + Hib as a booster.
* Subjects who received DTPw-HBV/Hib in the primary vaccination with HBV at birth will receive DTPw-HBV/Hib vaccine as a booster.

ELIGIBILITY:
Inclusion criteria:

For subjects receiving Plain PRP followed by DTPw-HBV:

Male or female infant, 10 to 11 months of age, who previously completed the three-dose primary vaccination course with the DTPw-HBV/Hib vaccine.

For subjects receiving DTPw-HBV/Hib or DTPw-HBV + Hib:

Male or female infant, 15-18 months of age, who previously completed the three-dose primary vaccination course with the DTPw-HBV/Hib vaccine.

For all subjects:

* Subjects who the investigator believes that their parent/guardian can and will comply with the requirements of the protocol.
* Free of obvious health problems as established by medical history and clinical examination

Exclusion criteria:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding administration of the study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to administration of the study vaccine.
* Planned administration/administration of a vaccine not foreseen by the study protocol starting 30 days before and ending 30 days after administration of the study vaccine with the exception of oral polio vaccine.

Ages: 10 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 745 (Actual)
Dates: Start 2005-02-10 (Actual); Primary Completion 2006-03-01 (Actual); Study Completion 2006-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Philippines (3):
  - GSK Investigational Site, City of Muntinlupa
  - GSK Investigational Site, Pasay
  - GSK Investigational Site, Quezon City

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Gatchalian et al. A new DTPw-HBV/Hib vaccine: Immunogenic and safe for primary vaccination and booster dosing in the second year of life - 5th World Congress WSPID, Bangkok, Thailand, 15-18 Nov 2007
- [Background] Gatchalian S, Reyes M, Bermal N, Chandrasekaran V, Han HH, Bock HL, Lefevre I. A new DTPw-HBV/Hib vaccine: immune memory after primary vaccination and booster dosing in the second year of life. Hum Vaccin. 2008 Jan-Feb;4(1):60-6. doi: 10.4161/hv.4.1.5069. Epub 2007 Sep 23. PMID 18376148
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 104065 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104065 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104065 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104065 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104065 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104065 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Tritanrix-HepB/Hiberix Kft. Mix Group: Healthy male and female infants who were primed with Tritanrix-HepB/Hiberix Kft. vaccine, received a booster dose of Tritanrix-HepB/Hiberix Kft. administered intramuscularly into the right upper thigh, at 15-18 months of age.
- Tritanrix-HepB/Hiberix Kft. Ref Group: Healthy male and female infants who were primed with Tritanrix-HepB/Hiberix vaccine, received a booster dose of Tritanrix-HepB/Hiberix Kft. administered intramuscularly into the right upper thigh, at 15-18 months of age.
- HB Tritanrix-HepB/Hiberix Kft. Mix Group: Healthy male and female infants who were primed with Tritanrix-HepB/Hiberix Kft. vaccine (with HepB at birth), received a booster dose of Tritanrix-HepB/Hiberix Kft. administered intramuscularly into the right upper thigh, at 15-18 months of age.
- Tritanrix-HepB Kft.+Hiberix Group: Healthy male and female infants who were primed with Tritanrix-HepB Kft. and Hiberix vaccines, were boosted with Tritanrix-HepB Kft. vaccine administered intramuscularly into the right upper thigh and Hiberix vaccine, administered intramuscularly into the left upper thigh, at 15-18 months of age.
- PRP Tritanrix-HepB Kft. Mix Group: Healthy male and female infants who were primed with Tritanrix-HepB/Hiberix Kft. vaccine, received plain Polyribosil-Ribitol-Phosphate (PRP) polysaccharide vaccine administered intramuscularly into the right upper thigh, at 10 months of age, followed by a booster dose of Tritanrix-HepB Kft. administered intramuscularly into the right upper thigh, at 15-18 months of age.
- PRP Tritanrix-HepB Kft. Ref Group: Healthy male and female infants who were primed with Tritanrix-HepB/Hiberix vaccine, received plain Polyribosil-Ribitol-Phosphate (PRP) polysaccharide vaccine administered intramuscularly into the right upper thigh, at 10 months of age, followed by a booster dose of Tritanrix-HepB Kft. administered intramuscularly into the right upper thigh, at 15-18 months of age.
Period: Overall Study
Arm/Group | Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB/Hiberix Kft. Ref Group | HB Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB Kft.+Hiberix Group | PRP Tritanrix-HepB Kft. Mix Group | PRP Tritanrix-HepB Kft. Ref Group
Started | 119 | 124 | 167 | 250 | 42 | 43
Completed | 119 | 123 | 166 | 250 | 41 | 41
Not Completed | 0 | 1 | 1 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Migrated/moved from study area | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to follow-up (incompl. vaccination) | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to follow-up (compl. vaccination) | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PRP Tritanrix-HepB Kft. Mix Group: Healthy male and female infants who were primed with Tritanrix-HepB/Hiberix Kft. vaccine, received plain PRP polysaccharide vaccine administered intramuscularly into the right upper thigh, at 10 months of age, followed by a booster dose of Tritanrix-HepB Kft. administered intramuscularly into the right upper thigh, at 15-18 months of age.
- PRP Tritanrix-HepB Kft. Ref Group: Healthy male and female infants who were primed with Tritanrix-HepB/Hiberix vaccine, received plain PRP polysaccharide vaccine administered intramuscularly into the right upper thigh, at 10 months of age, followed by a booster dose of Tritanrix-HepB Kft. administered intramuscularly into the right upper thigh, at 15-18 months of age.
- Total: Total of all reporting groups
Arm/Group | Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB/Hiberix Kft. Ref Group | HB Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB Kft.+Hiberix Group | PRP Tritanrix-HepB Kft. Mix Group | PRP Tritanrix-HepB Kft. Ref Group | Total
Number analyzed (Participants) | 119 | 124 | 167 | 250 | 42 | 43 | 745
Age, Continuous [Mean (Standard Deviation); unit: Months] | 14.5 (1.44) | 14.8 (2.07) | 14.7 (1.89) | 15.0 (2.04) | 9.9 (0.68) | 9.8 (0.61) | 14.23 (1.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 58 | 90 | 120 | 21 | 21 | 359
  Male | 70 | 66 | 77 | 130 | 21 | 22 | 386
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  East/South East Asian heritage | 119 | 124 | 167 | 250 | 42 | 43 | 745

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-PRP Antibody Concentrations ≥ 0.15 μg/mL and ≥ 1.0 μg/mL
Description: The number of subjects with anti-PRP antibody concentrations equal to or above (≥) 0.15 μg/mL and ≥ 1.0 μg/mL, at one month after the PRP challenge.
Time Frame: At Month 1, post-PRP challenge
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | PRP Tritanrix-HepB Kft. Mix Group | PRP Tritanrix-HepB Kft. Ref Group
Number analyzed (Participants) | 39 | 41
Participants
  Anti-PRP ≥ 0.15 μg/mL | 39 | 41
  Anti-PRP ≥ 1.0 μg/mL | 37 | 39

2. Primary Outcome: Number of Subjects With Anti-PRP Antibody Concentrations ≥ 0.15 μg/mL and ≥ 1.0 μg/mL.
Description: The number of subjects with anti-PRP antibody concentrations equal to or above (≥) 0.15 μg/mL and ≥ 1.0 μg/mL, at one month post-booster vaccination.
Time Frame: At Month 1, post-booster vaccination
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB/Hiberix Kft. Ref Group | HB Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB Kft.+Hiberix Group
Number analyzed (Participants) | 77 | 71 | 88 | 74
Participants
  Anti-PRP ≥ 0.15 μg/mL | 77 | 71 | 88 | 74
  Anti-PRP ≥ 1.0 μg/mL | 76 | 70 | 88 | 74

3. Primary Outcome: Number of Seroprotected Subjects Against Diphteria (D) and Tetanus (T)
Description: A seroprotected subject was defined as a vaccinated subject, with anti-D and anti-T antibody concentrations equal to or above (≥) 0.1 International Units per milliliter (IU/mL).
Time Frame: At Month 1, post-booster vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB/Hiberix Kft. Ref Group | HB Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB Kft.+Hiberix Group
Number analyzed (Participants) | 77 | 71 | 88 | 74
Participants
  Anti-D: number analyzed (Participants) | 77 | 70 | 88 | 73
  Anti-D | 74 | 68 | 88 | 73
  Anti-T | 77 | 71 | 88 | 74

4. Primary Outcome: Seroprotection Rates for Anti-D Antibodies
Description: The seroprotection rate is defined as the estimated proportion of subjects with protective antibodies as assessed by the Enzyme-Linked Immunosorbent Assay (ELISA) (antibody concentration ≥ 0.1 IU/mL), or by Vero-cell neutralisation assay (antibody concentration ≥ 0.016 IU/mL), for subjects seronegative as assessed by ELISA.
Time Frame: At Month 1, post-booster vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Proportion
Arm/Group | Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB/Hiberix Kft. Ref Group | HB Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB Kft.+Hiberix Group
Number analyzed (Participants) | 77 | 70 | 88 | 73
Proportion | 100 [95.3 to 100] | 100 [94.9 to 100] | 100 [95.9 to 100] | 100 [95.1 to 100]

5. Primary Outcome: Number of Seroprotected Subjects Against Hepatitis B Surface Antigen (HBs)
Description: A seroprotected subject was defined as a vaccinated subject with an anti-HBs antibody concentration equal to or above (≥) 10 milli International Units per milliliter (mIU/mL).
Time Frame: At Month 1, post-booster vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB/Hiberix Kft. Ref Group | HB Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB Kft.+Hiberix Group
Number analyzed (Participants) | 77 | 71 | 88 | 74
Participants | 74 | 69 | 84 | 72

6. Primary Outcome: Number of Seroprotected Subjects Against Bordetella Pertussis (BPT)
Description: A seroprotected subject was defined as a vaccinated subject with an anti-BPT antibody concentration equal to or above (≥) 15 ELISA units per milliliter (EL.U/mL).
Time Frame: At Month 1, post-booster vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB/Hiberix Kft. Ref Group | HB Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB Kft.+Hiberix Group
Number analyzed (Participants) | 74 | 65 | 85 | 69
Participants | 74 | 65 | 85 | 69

7. Primary Outcome: Number of Subjects With Booster Response to BPT Antigen
Description: The booster response was defined as:
  * an anti-BPT antibody concentration equal to or above (≥) the cut-off value (15 EL.U/mL) at post-booster vaccination in subjects seronegative (anti-BPT antibody concentration < 15 EL.U/mL) prior to administration of the booster dose; or
  * at least a 2-fold increase in antibody concentration from pre- to post-vaccination time points, in subjects who were seropositive (anti-BPT antibody concentration ≥ 15 EL.U/mL) prior to the administration of the booster dose.
Time Frame: At Month 1, post-booster vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB/Hiberix Kft. Ref Group | HB Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB Kft.+Hiberix Group
Number analyzed (Participants) | 72 | 65 | 84 | 68
Participants | 70 | 64 | 79 | 67

8. Primary Outcome: Anti-PRP Antibody Concentrations
Description: Anti-PRP antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in microgram per milliliter (μg/mL), as assessed by ELISA.
Time Frame: At Month 1, post-PRP challenge
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | PRP Tritanrix-HepB Kft. Mix Group | PRP Tritanrix-HepB Kft. Ref Group
Number analyzed (Participants) | 39 | 41
μg/mL | 33.190 [18.546 to 59.397] | 22.727 [13.524 to 38.192]

9. Primary Outcome: Anti-PRP Antibody Concentrations.
Description: as for outcome 8
Time Frame: At Month 1, post-booster vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB/Hiberix Kft. Ref Group | HB Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB Kft.+Hiberix Group
Number analyzed (Participants) | 77 | 71 | 88 | 74
μg/mL | 56.670 [42.276 to 75.964] | 81.681 [58.576 to 113.900] | 58.669 [45.568 to 75.537] | 113.073 [82.280 to 155.389]

10. Primary Outcome: Anti-D and Anti-T Antibody Concentrations
Description: Anti-D and anti-T antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in International Units per milliliter (IU/mL), as assessed by ELISA.
Time Frame: At Month 1, post-booster vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB/Hiberix Kft. Ref Group | HB Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB Kft.+Hiberix Group
Number analyzed (Participants) | 77 | 71 | 88 | 74
IU/mL
  Anti-D: number analyzed (Participants) | 77 | 70 | 88 | 73
  Anti-D | 3.087 [2.206 to 4.319] | 1.812 [1.354 to 2.425] | 3.452 [2.692 to 4.425] | 3.128 [2.344 to 4.174]
  Anti-T | 13.371 [10.846 to 16.484] | 12.181 [9.994 to 14.848] | 12.838 [10.548 to 15.626] | 16.822 [13.682 to 20.682]

11. Primary Outcome: Anti-HBs Antibody Concentrations
Description: Anti-HBs antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in milli International Units per milliliter (mIU/mL), as assessed by ELISA.
Time Frame: At Month 1, post-booster vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB/Hiberix Kft. Ref Group | HB Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB Kft.+Hiberix Group
Number analyzed (Participants) | 77 | 71 | 88 | 74
mIU/mL | 2400.0 [1399.5 to 4115.8] | 1628.3 [1041.4 to 2546.0] | 2467.9 [1554.2 to 3918.9] | 2465.1 [1572.6 to 3864.2]

12. Primary Outcome: Anti-BPT Antibody Concentrations
Description: Anti-BPT antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in ELISA units per milliliter (EL.U/mL), as assessed by ELISA.
Time Frame: At Month 1, post-booster vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB/Hiberix Kft. Ref Group | HB Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB Kft.+Hiberix Group
Number analyzed (Participants) | 74 | 65 | 85 | 69
EL.U/mL | 91.3 [82.1 to 101.4] | 118.8 [105.0 to 134.4] | 97.6 [89.0 to 107.1] | 93.5 [82.4 to 106.0]

13. Secondary Outcome: Number of Subjects With Anti-PRP Antibody Concentrations ≥ 0.15 μg/mL and ≥ 1.0 μg/mL
Description: The number of subjects with anti-PRP antibody concentrations equal to or above (≥) 0.15 μg/mL and ≥ 1.0 μg/mL, prior to the PRP challenge.
Time Frame: At Month 0, prior to the PRP challenge
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PRP Tritanrix-HepB Kft. Mix Group | PRP Tritanrix-HepB Kft. Ref Group
Number analyzed (Participants) | 38 | 41
Participants
  Anti-PRP ≥ 0.15 μg/mL | 37 | 41
  Anti-PRP ≥ 1.0 μg/mL | 32 | 34

14. Secondary Outcome: Number of Subjects With Anti-PRP Antibody Concentrations ≥ 0.15 μg/mL and ≥ 1.0 μg/mL.
Description: The number of subjects with anti-PRP antibody concentrations equal to or above (≥) 0.15 μg/mL and ≥ 1.0 μg/mL, prior to the booster vaccination.
Time Frame: At Month 0, prior to the PRP challenge
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB/Hiberix Kft. Ref Group | HB Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB Kft.+Hiberix Group
Number analyzed (Participants) | 77 | 71 | 89 | 74
Participants
  Anti-PRP ≥ 0.15 μg/mL | 74 | 69 | 84 | 72
  Anti-PRP ≥ 1.0 μg/mL | 53 | 62 | 66 | 49

15. Secondary Outcome: Number of Subjects With Anti-D and Anti-T Antibody Concentrations ≥ the Cut-off Value
Description: The number of subjects with anti-D antibody concentrations equal to or above (≥) the cut-off value of 0.1 IU/mL as assessed by ELISA, (or ≥ 0.016 IU/mL as assessed by the neutralisation assay on Vero cells in subjects seronegative by ELISA testing) and, the number of subjects with anti-T antibody concentrations ≥ the cut-off value of 0.1 IU/mL as assessed by ELISA.
Time Frame: At Month 0, prior to the PRP challenge
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB/Hiberix Kft. Ref Group | HB Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB Kft.+Hiberix Group
Number analyzed (Participants) | 77 | 72 | 89 | 74
Participants
  Anti-D | 45 | 24 | 58 | 46
  Anti-T | 72 | 67 | 86 | 69

16. Secondary Outcome: Seroprotection Rates for Anti-D Antibodies
Description: The seroprotection rate is defined as the estimated proportion of subjects with protective antibodies as assessed by ELISA (antibody concentration ≥ 0.1 IU/mL), or by Vero-cell neutralisation assay (antibody concentration ≥ 0.016 IU/mL), for subjects seronegative as assessed by ELISA.
Time Frame: At Month 0, prior to the PRP challenge
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Proportion
Arm/Group | Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB/Hiberix Kft. Ref Group | HB Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB Kft.+Hiberix Group
Number analyzed (Participants) | 77 | 72 | 89 | 74
Proportion | 85.7 [75.9 to 92.6] | 71.6 [61.1 to 82.1] | 95.5 [88.9 to 98.8] | 85.1 [75.0 to 92.3]

17. Secondary Outcome: Number of Subjects With Anti-HBs Antibody Concentrations ≥ the Cut-off Value
Description: The number of subjects with anti-HBs antibody concentrations equal to or above (≥) the cut-off value of 10 mIU/mL, prior to the booster vaccination.
Time Frame: At Month 0, prior to the PRP challenge
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB/Hiberix Kft. Ref Group | HB Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB Kft.+Hiberix Group
Number analyzed (Participants) | 77 | 72 | 89 | 74
Participants | 56 | 44 | 69 | 56

18. Secondary Outcome: Number of Subjects With Anti-BPT Antibody Concentrations ≥ the Cut-off Value
Description: The number of subjects with anti-BPT antibody concentrations equal to or above (≥) the cut-off value of 15 EL.U/mL, prior to the booster vaccination.
Time Frame: At Month 0, prior to the PRP challenge
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB/Hiberix Kft. Ref Group | HB Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB Kft.+Hiberix Group
Number analyzed (Participants) | 75 | 72 | 88 | 73
Participants | 23 | 21 | 33 | 27

19. Secondary Outcome: Anti- PRP Antibody Concentrations
Description: as for outcome 8
Time Frame: At Month 0, prior to the PRP challenge
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | PRP Tritanrix-HepB Kft. Mix Group | PRP Tritanrix-HepB Kft. Ref Group
Number analyzed (Participants) | 38 | 41
μg/mL | 4.683 [2.602 to 8.428] | 4.507 [2.914 to 6.971]

20. Secondary Outcome: Anti- PRP Antibody Concentrations.
Description: as for outcome 8
Time Frame: At Month 0, prior to the PRP challenge
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB/Hiberix Kft. Ref Group | HB Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB Kft.+Hiberix Group
Number analyzed (Participants) | 77 | 71 | 89 | 74
μg/mL | 2.703 [1.771 to 4.125] | 5.312 [3.496 to 8.070] | 2.837 [1.953 to 4.121] | 2.904 [1.905 to 4.426]

21. Secondary Outcome: Anti-D and Anti-T Antibody Concentrations.
Description: as for outcome 10
Time Frame: At Month 0, prior to the PRP challenge
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB/Hiberix Kft. Ref Group | HB Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB Kft.+Hiberix Group
Number analyzed (Participants) | 77 | 72 | 89 | 74
IU/mL
  Anti-D | 0.117 [0.097 to 0.141] | 0.077 [0.066 to 0.090] | 0.162 [0.127 to 0.206] | 0.145 [0.116 to 0.181]
  Anti-T | 0.397 [0.321 to 0.491] | 0.512 [0.400 to 0.656] | 0.588 [0.464 to 0.745] | 0.446 [0.353 to 0.564]

22. Secondary Outcome: Anti-HBs Antibody Concentrations.
Description: as for outcome 11
Time Frame: At Month 0, prior to the PRP challenge
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB/Hiberix Kft. Ref Group | HB Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB Kft.+Hiberix Group
Number analyzed (Participants) | 77 | 72 | 89 | 74
mIU/mL | 43.6 [29.4 to 64.8] | 26.1 [18.0 to 38.0] | 70.5 [46.9 to 105.8] | 43.6 [29.8 to 63.7]

23. Secondary Outcome: Anti-BPT Antibody Concentrations.
Description: as for outcome 12
Time Frame: At Month 0, prior to the PRP challenge
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB/Hiberix Kft. Ref Group | HB Tritanrix-HepB/Hiberix Kft. Mix Group | Tritanrix-HepB Kft.+Hiberix Group
Number analyzed (Participants) | 75 | 72 | 88 | 73
EL.U/mL | 10.6 [9.4 to 12.1] | 10.7 [9.3 to 12.2] | 12.8 [10.9 to 15.1] | 11.9 [10.3 to 13.8]

24. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 20 millimeters (mm) of injection site.
Time Frame: During the 4-Day (Days 0-3) post-PRP challenge
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one vaccine administration documented and with the symptoms sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | PRP Tritanrix-HepB Kft. Mix Group | PRP Tritanrix-HepB Kft. Ref Group
Number analyzed (Participants) | 41 | 42
Participants
  Any Pain | 13 | 12
  Grade 3 Pain | 0 | 0
  Any Redness | 11 | 15
  Grade 3 Redness | 0 | 0
  Any Swelling | 7 | 11
  Grade 3 Swelling | 0 | 0

25. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)], irritability and loss of appetite. Any = occurrence of the symptom regardless of intensity grade. Grade 3 drowsiness = drowsiness that prevented normal activity. Grade 3 fever = fever > 39.5 °C. Grade 3 irritability = crying that could not be comforted and prevented normal activity. Grade 3 loss of appetite = not eating at all. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 4-Day (Days 0-3) post-PRP challenge
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | PRP Tritanrix-HepB Kft. Mix Group | PRP Tritanrix-HepB Kft. Ref Group
Number analyzed (Participants) | 41 | 42
Participants
  Any Drowsiness | 6 | 10
  Grade 3 Drowsiness | 0 | 0
  Related Drowsiness | 6 | 10
  Any Fever (Axillary) | 4 | 7
  Grade 3 Fever (Axillary) | 0 | 0
  Related Fever (Axillary) | 4 | 7
  Any Irritability | 11 | 8
  Grade 3 Irritability | 0 | 0
  Related Irritability | 11 | 8
  Any Loss of appetite | 5 | 7
  Grade 3 Loss of appetite | 0 | 0
  Related Loss of appetite | 5 | 7

26. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms.
Description: as for outcome 24
Time Frame: During the 4-Day (Days 0-3) post-booster vaccination period
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Groups:
- PRP Pooled Group: PRP Tritanrix-HepB Kft. Mix Group and PRP Tritanrix-HepB Kft. Ref Group were pooled into PRP Pooled Group.
- Mix Pooled Group: Tritanrix-HepB/Hiberix Kft. Mix Group, HB Tritanrix-HepB/Hiberix Kft. Mix Group and Tritanrix-HepB/Hiberix Kft. Ref Group were pooled into Mix Pooled Group.
Arm/Group | PRP Pooled Group | Mix Pooled Group | Tritanrix-HepB Kft.+Hiberix Group
Number analyzed (Participants) | 82 | 409 | 250
Participants
  Any Pain | 56 | 303 | 181
  Grade 3 Pain | 11 | 57 | 34
  Any Redness | 46 | 255 | 152
  Grade 3 Redness | 7 | 58 | 50
  Any Swelling | 44 | 250 | 140
  Grade 3 Swelling | 16 | 84 | 65

27. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms.
Description: as for outcome 25
Time Frame: During the 4-Day (Days 0-3) post-booster vaccination period
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | PRP Pooled Group | Mix Pooled Group | Tritanrix-HepB Kft.+Hiberix Group
Number analyzed (Participants) | 82 | 409 | 250
Participants
  Any Drowsiness | 34 | 174 | 105
  Grade 3 Drowsiness | 1 | 11 | 4
  Related Drowsiness | 33 | 174 | 104
  Any Fever (Axillary) | 59 | 270 | 168
  Grade 3 Fever (Axillary) | 2 | 10 | 1
  Related Fever (Axillary) | 59 | 270 | 168
  Any Irritability | 54 | 267 | 162
  Grade 3 Irritability | 2 | 17 | 11
  Related Irritability | 54 | 266 | 161
  Any Loss of appetite | 25 | 129 | 79
  Grade 3 Loss of appetite | 1 | 6 | 1
  Related Loss of appetite | 25 | 129 | 79

28. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-Day (Day 0-30) follow-up period
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | PRP Pooled Group | Mix Pooled Group | Tritanrix-HepB Kft.+Hiberix Group
Number analyzed (Participants) | 85 | 410 | 250
Participants | 22 | 27 | 14

29. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Month 0 to Month 9.5)
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | PRP Pooled Group | Mix Pooled Group | Tritanrix-HepB Kft.+Hiberix Group
Number analyzed (Participants) | 85 | 410 | 250
Participants | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-Day (Day 0-3) post-vaccination period (PRP challenge and booster); Unsolicited AEs: during the 31-Day (Day 0-30) post-booster; SAEs: during the entire study period (from Month 0 up to Month 9.5).
Groups:
- PRP TRITANRIX-HEPB KFT. MIX GROUP: Healthy male and female infants who were primed with Tritanrix -HepB/Hiberix Kft. vaccine, received plain PRP polysaccharide vaccine administered intramuscularly into the right upper thigh, at 10 months of age, followed by a booster dose of Tritanrix-HepB Kft. administered intramuscularly into the right upper thigh, at 15-18 months of age .
- PRP TRITANRIX-HEPB KFT. REF GROUP: Healthy male and female infants who were primed with Tritanrix -HepB/Hiberix vaccine, received plain PRP polysaccharide vaccine administered intramuscularly into the right upper thigh, at 10 months of age, followed by a booster dose of Tritanrix-HepB Kft. administered intramuscularly into the right upper thigh, at 15-18 months of age .
Arm/Group | PRP Pooled Group | Mix Pooled Group | Tritanrix-HepB Kft.+Hiberix Group | PRP TRITANRIX-HEPB KFT. MIX GROUP | PRP TRITANRIX-HEPB KFT. REF GROUP
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/410 | 0/250 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/85 | 0/410 | 0/250 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 77/85 | 379/410 | 231/250 | 37/42 | 40/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PRP Pooled Group (N=85) | Mix Pooled Group (N=410) | Tritanrix-HepB Kft.+Hiberix Group (N=250) | PRP TRITANRIX-HEPB KFT. MIX GROUP (N=0) | PRP TRITANRIX-HEPB KFT. REF GROUP (N=0)
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | PRP Pooled Group (N=85) | Mix Pooled Group (N=410) | Tritanrix-HepB Kft.+Hiberix Group (N=250) | PRP TRITANRIX-HEPB KFT. MIX GROUP (N=42) | PRP TRITANRIX-HEPB KFT. REF GROUP (N=43)
Upper respiratory tract infection (Infections and infestations) | 8 | 8 | 8 | 0 | 0
Pain (post-booster) (General disorders) | 56/82 | 303/409 | 181 | 0 | 0
Redness (post-booster) (General disorders) | 46/82 | 255/409 | 152 | 0 | 0
Swelling (post-booster) (General disorders) | 44/82 | 250/409 | 140 | 0 | 0
Drowsiness (post-booster) (General disorders) | 34/82 | 174/409 | 105 | 0 | 0
Fever (Axillary) (post-booster) (General disorders) | 59/82 | 270/409 | 168 | 0 | 0
Iritability (post-booster) (General disorders) | 54/82 | 267/409 | 162 | 0 | 0
Loss of appetite (post-booster) (General disorders) | 25/82 | 129/409 | 79 | 0 | 0
Pain (post-PRP challenge) (General disorders) | 0/0 | 0/0 | 0/0 | 13 | 12
Redness (post-PRP challenge) (General disorders) | 0/0 | 0/0 | 0/0 | 11 | 15
Swelling (post-PRP challenge) (General disorders) | 0/0 | 0/0 | 0/0 | 7 | 11
Drowsiness (post-PRP challenge) (General disorders) | 0/0 | 0/0 | 0/0 | 6 | 10
Fever (Axillary) (post-PRP challenge) (General disorders) | 0/0 | 0/0 | 0/0 | 4 | 7
Irritability (post-PRP challenge) (General disorders) | 0/0 | 0/0 | 0/0 | 11 | 8
Loss of appetite (post-PRP challenge) (General disorders) | 0/0 | 0/0 | 0/0 | 5 | 7

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.